CLINICAL TRIAL: NCT04980807
Title: An Open Observational Study of Clinical and Electrophysiological Outcomes in Male and Female Patients With CMT Type 1 & 2, and Aged-matched Healthy Controls
Brief Title: Observational Study of Neuromuscular Function in CMT Type 1&2 and Healthy Controls
Acronym: ESTABLISH
Status: Completed | Type: Observational
Sponsor: NMD Pharma A/S (Industry)
Collaborators: Aarhus University Hospital (Other); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: CMT Observational
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-07

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: Neuromuscular Junction Transmission; Repetitive Nerve Stimulation; Neuromuscular Disease; Single Fiber EMG
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMT Patients: Individuals with Charcot-Marie-Tooth Disease Types 1 and 2.
- Healthy Controls: Healthy age-matched volunteers

SUMMARY:
The primary aim of this study is to discover whether patients with CMT type 1 and 2 have neuromuscular junction transmission deficits.

The secondary aim is to collect information of different clinical and electrophysiological test procedures to perform possible future clinical trials in CMT patients.

DETAILED DESCRIPTION:
The study is a prospective observational pilot study involving two investigational sites:

1. Department of Neurology, Arhus University Hospital
2. Department of Neurology, Ohio State University

A total of 20 patients with Charcot-Marie-Tooth (CMT) disease and 10 healthy age-matched controls will be included with each site including 10 CMT patients and 5 Healthy Controls. CMT patients will undergo electrophysiological (repetitive nerve stimulation and single fiber EMG analyses) and functional (different tests of muscle strength, fatigability, dexterity, and balance) testing on 4 separate occasions. Healthy controls will undergo electrophysiological testing at baseline only.

To assess whether patients with CMT have deficits in NMJ transmission, results from repetitive nerve stimulation and single fiber EMG analyses in CMT patients will be compared to those obtained in healthy controls at baseline. To inform future clinical trials, results relability and tolerability estimates obtained from sequential electrophysiological and functional tests will be calculated

ELIGIBILITY:
Inclusion Criteria for CMT Patients

* Age ≥ 18 years
* Diagnosis of CMT confirmed by:
* Clinical presentation and electro diagnostics or genetics
* Physical Features (all must apply): 1) Ambulation for at least 10 meters, without a brace 2) Left and right ankle plantar flexion Medical Research Council (MRC) grade 2 to 5, inclusive 3) Left and right ankle dorsiflexion MRC manual muscle testing (MMT) grade 2 to 4+, inclusive.
* Ability to adhere to the study visit schedule/procedures, and to understand and comply with protocol requirements
* Stable concomitant medications for 2 months prior to enrolment
* Signed written informed consent

Exclusion Criteria for CMT Patients

* Severe deformity or ankle contracture that would sufficiently limit passive range of motion to affect assessment of dorsiflexion strength
* Ulceration that would interfere with functional ability
* Recent major surgery
* Significant change in physical activity or exercise (e.g., significant increase or decrease in intensity or frequency) within 8 weeks before Study Day 1 or inability to maintain the baseline level of physical activity throughout the study
* Any disability or condition that would prevent completion of the study tasks
* Moderate to severe Neuropathic or inflammatory/musculoskeletal pain that would interfere with performance of the tests
* A diagnosis of a primary NMJ disorder such as myasthenia gravis, Lambert Eaton Myasthenic Syndrome or congenital myasthenic disorder

Inclusion Criteria for Healthy Volunteers

* Healthy male or female volunteers
* Age ≥18 years
* Able to give written informed consent

Exclusion Criteria for Healthy Volunteers

* Pregnant
* Requiring prescription medicines likely to interfere with electromyography (EMG) recordings
* Presence of current or previous medical condition which might interfere with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible CMT patients will be invited to participate at the respective study sites. Age matched healthy volunteers will be recruited through advertisement at the respective study sites
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Repetitive Nerve Stimulation - difference between CMT patients and healthy controls | Baseline
  Percentage decrement of CMAP for the trapezius
Repetitive Nerve Stimulation - difference between CMT patients and healthy controls | Baseline
  Percentage decrement of CMAP for abductor pollicis brevis
Single Fiber Electro Myography (sfEMG) - difference between CMT patients and healthy controls | Baseline
  Percentage blocking
Single Fiber Electro Myography (sfEMG) - difference between CMT patients and healthy controls | Baseline
  Jitter

SECONDARY OUTCOMES:
Isometric Dynamometry - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test will be used to evaluate maximum isometric strength
Manual Muscle Testing - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test is a physical examination of muscle strength. 15 muscle groups/motions will be tested. 13 of these are tested bilaterally. A total score between (0-280) is calculated
9 Hole Peg Test - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This is a test of finger dexterity
6-Spot Step Test - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test is a quantitative measure of lower extremity function
10-Meter Walk/run Test - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test measures how fast the participant can walk/run 10 meters.
Timed Up and Go - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test measures how fast the participant can stand from a chair, walk 3 meters, turn around, return, and sit in the chair at a comfortable and safe pace
Berg Balance Scale - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  The test measures balance during different functional tasks. A total score is calculated as the sum of the individual scores for each item, with maximum value 56, with a lower score meaning worse balance
6 Minute Walk Test - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  This test measures how far a person can walk in six minutes
Single Fiber Electro Myography (sfEMG) - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  Percantage blocking
Single Fiber Electro Myography (sfEMG) - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  Jitter
Repetitive Nerve Stimulation - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  Percentage decrement of CMAP for Trapezius
Repetitive Nerve Stimulation - test reliability in patients with CMT | The test is performed at baseline and day 14, 28 and 42.
  Percentage decrement of CMAP for abductor pollicis brevis

OTHER OUTCOMES:
CMTES2 Score | This test is performed at baseline in individuals with CMT disease
  This test measures CMT disease severity. Total score is calculated as the sum of the 7 sub-scores with a maximum of score of 28
Adverse Events | At baseline for healthy controls and from baseline until final visit at day 42 for CMT patients
  Number of adverse events by severity
Tolerability of test procedures | Performed for each test at each visit (baseline, day 14, 28 and 42)
  The tolerability score assessed on a 0-9 rating scale (0=no discomfort to 9=worst possible discomfort)
Association between NMJ function and clinical function in CMT patients | Baseline
  Correlation

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD, PhD, Principal Investigator — Aarhus University Hospital; William D Arnold, MD, Principal Investigator — Ohio State University
Locations (2):
- Ohio State University, Columbus, Ohio, United States
- Aarhus University Hospital, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No